CLINICAL TRIAL: NCT05367687
Title: A Randomized, Open-Label, Multi-Center, Phase 2 Clinical Study of Camrelizumab Plus Rivoceranib (Apatinib) Versus Camrelizumab as Adjuvant Therapy in Patients With Hepatocellular Carcinoma (HCC) at High Risk of Recurrence After Curative Resection or Ablation
Brief Title: A Study to Evaluate Camrelizumab Plus Rivoceranib (Apatinib) Versus Camrelizumab as Adjuvant Therapy in Patients With Hepatocellular Carcinoma (HCC) at High Risk of Recurrence After Curative Resection or Ablation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHR-1210-II-218
Record Dates: First submitted 2022-05-06; First posted 2022-05-10 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Adjuvant Therapy in Patients With Hepatocellular Carcinoma (HCC) at High Risk of Recurrence After Curative Resection or Ablation
MeSH Terms: interventions — camrelizumab

STUDY DESIGN:
Masking Description: Camrelizumab Plus Rivoceranib (Apatinib) compared with Camrelizumab
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Experimental): Camrelizumab Plus Rivoceranib (Apatinib)
  Interventions: Drug: Camrelizumab、Rivoceranib
- Control group (Active Comparator): Camrelizumab
  Interventions: Drug: Camrelizumab

INTERVENTIONS:
Drug: Camrelizumab、Rivoceranib — Camrelizumab: 200 mg, intravenous infusion. Rivoceranib: 250 mg, oral.
  Arms: Treatment group
Drug: Camrelizumab — Camrelizumab: 200 mg, intravenous infusion.
  Arms: Control group

SUMMARY:
A Trial to Evaluate the Efficacy and Safety of Camrelizumab Plus Rivoceranib (Apatinib) Versus Camrelizumab as Adjuvant Therapy in Patients with Hepatocellular Carcinoma (HCC) at High Risk of Recurrence After Curative Resection or Ablation.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects with a histopathological diagnosis of HCC.
2. Subjects who have undergone a curative resection or ablation (radiofrequency ablation [RFA] or microwave ablation [MVA] only).
3. No previous systematic treatment and locoregional therapy for HCC prior to randomization.
4. Absence of major macrovascular invasion.
5. No extrahepatic spread.
6. Full recovery from Curative resection or ablation within 4 weeks prior to randomization.
7. High risk for HCC recurrence after resection or ablation.
8. For patients who received post-operative transarterial chemoembolization: full recovery from the procedure within 4 weeks prior to randomization.
9. Child-Pugh Class: Grade A.
10. ECOG-PS score: 0 or 1.
11. Subjects with HCV- RNA (+) must receive antiviral therapy.
12. Adequate organ function.

Exclusion Criteria:

1. Known hepatocholangiocarcinoma, sarcomatoid HCC, mixed cell carcinoma and fibrolamellar HCC; other active malignant tumor except HCC within 5 years or simultaneously.
2. Evidence of residual lesion, recurrence, and metastasis at randomization.
3. Moderate-to-severe ascites with clinical symptoms.
4. History of hepatic encephalopathy.
5. History of gastrointestinal hemorrhage within 6 months prior to the start of study treatment or clear tendency of gastrointestinal haemorrhage.
6. Active or history of autoimmune disease.
7. Interstitial lung disease that is symptomatic or may interfere with the detection and management of suspected drug-related pulmonary toxicity.
8. Cardiac clinical symptom or cardiovascular disease that is not well controlled.
9. Severe infection within 4 weeks prior to the start of study treatment.
10. Subjects with inadequately controlled hypertension or history of hypertensive crisis or hypertensive encephalopathy.
11. Thrombosis or thromboembolic event within 6 months prior to the start of study treatment.
12. Known genetic or acquired hemorrhage or thrombotic tendency.
13. Previous or current presence of metastasis to central nervous system.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 251 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2024-11-15 (Actual); Study Completion 2024-11-15 (Actual)

PRIMARY OUTCOMES:
Recurrence-Free Survival (RFS), as Determined by the investigator | Randomization up to approximately 43 months
  RFS is defined as the time from randomization to the first documented occurrence of local, regional, or metastatic HCC as determined by the investigator, or death from any cause (whichever occurs first).

SECONDARY OUTCOMES:
RFS Rate at 24 and 36 Months, as Assessed by the Investigator | Randomization up to 24 months and up to 36 months
Time to Recurrence (TTR) as determined by the investigator | Randomization up to approximately 43 months
  TTR defined as the time from randomization to first documented occurrence of local, regional, or metastatic HCC.
Overall Survival (OS) | Randomization up to approximately 43 months
  OS is defined as the time from randomization to death from any cause.
The incidence and severity of adverse events (AEs) and serious adverse events (SAEs) as assessed by CTCAE v5.0 | Randomization up to approximately 43 months

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Hospital, Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided